CLINICAL TRIAL: NCT03730116
Title: Multicenter Observational Open Program. Assessment of the Efficacy and Tolerability of the Fixed-dose Combination of Bisoprolol/Perindopril in Patients With Arterial Hypertension and Stable CAD in Daily Clinical Practice (STYLE)
Brief Title: Assessment of the Efficacy and Tolerability of the Fixed-dose Combination of Bisoprolol/Perindopril
Acronym: STYLE
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-05150-056-RUS
Record Dates: First submitted 2018-10-22; First posted 2018-11-05 (Actual); Results first posted 2020-12-23 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-11

CONDITIONS: Arterial Hypertension; CHD - Coronary Heart Disease
MeSH Terms: conditions — Hypertension; Coronary Artery Disease | interventions — Bisoprolol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the patients with HT and concomitant stable CAD
  Interventions: Drug: bisoprolol/perindopril FDC

INTERVENTIONS:
Drug: bisoprolol/perindopril FDC — the first and only single-pill combination of beta-blocker and ACE inhibitor

SUMMARY:
Study objective - to assess the efficacy, tolerability and adherence of bisoprolol/perindopril FDC in patients with HT and stable CAD in everyday practice.

Type of the program: multicenter, observational, uncontrolled, open program. The program will involve 480 general practitioners (GPs) and cardiologists from the primary care facilities.Each doctor includes four patients. It is planned to include not less than 1920 patients in total.

DETAILED DESCRIPTION:
Multicenter observational open program. Assessment of the efficacy and tolerability of the fixed-dose combination of bisoprolol/perindopril in patients with arterial hypertension and stable CAD in daily clinical practice (STYLE)

Study objectives and purposes:

Primary endpoints:

* efficacy of bisoprolol/perindopril FDC in patients with HT and stable CAD in everyday practice regarding the BP
* efficacy of bisoprolol/perindopril FDC in patients with HT and stable CAD in everyday practice regarding the angina

Secondary endpoints:

* impact on the quality of life of bisoprolol/perindopril FDC in patients with HT and stable CAD in everyday practice
* adherence to bisoprolol/perindopril FDC therapy in patients with HT and stable CAD in everyday practice The program will involve 480 general practitioners (GPs) and cardiologists from the primary care facilities. Each doctor includes four patients. It is planned to include not less than 1920 patients in total.

Milestones of the program:

FSI - November, 2018 LSLV- January, 2019 Database Lock - February, 2019 Statistic Report- May, 2019 Clinical Study Report- January, 2020

ELIGIBILITY:
Inclusion Criteria:

* Stable CAD, defined as stable angina pectoris of class 1-3 by CCS (Canadian Cardiovascular Society) classification;
* Previously or newly diagnosed essential hypertension
* Age 18 to 79 years old;
* Informed consent of the patient for participation in the program;
* Decision of the doctor to prescribe bisoprolol/perindopril FDC before the inclusion in the program in accordance to the instruction for use.

Exclusion Criteria:

* Stable angina pectoris, class 4;
* History of myocardial infarction or cerebrovascular event within the past 3 months;
* Unstable angina within the past 6 months;
* Chronic heart failure classes 3-4 (NYHA);
* Type 1 diabetes mellitus or decompensated type 2 diabetes mellitus;
* Any serious decompensated concomitant diseases requiring the regular medical therapy;
* Inability to understand the essence of the program and follow the recommendations;
* Contraindications to beta-blockers or ACE inhibitors using;
* Participation of the patient in other trials in the present time or within 30 days before the start of observational program.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to include into the program the patients with HT and concomitant stable CAD. It is planned to include not less than 1920 patients in total.
  The patient is included in the program, if the doctor decides to prescribe FDC with beta-blocker bisoprolol and ACE inhibitor perindopril in accordance to the instruction for use.
Sampling Method: Non-Probability Sample
Enrollment: 1909 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Boytsov, Study Chair
Locations (1):
- FSBI NMIC of Cardiology of the Ministry of Health of Russia, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
The sponsor reserves the exclusive right to all materials, information, unpublished documentation, results and information obtained during the research. The Sponsor reserves the right to send research data to the health authorities (individual registration cards, analysis results, reports).
  No unpublished documentation or information transmitted to researchers can be transferred to unauthorized persons without the prior written consent of Sponsor.

REFERENCES:
- [Derived] Boytsov SA, Burtsev YP, Khomitskaya YV, Karpov YA; STYLE study investigators. Effectiveness and Tolerability of the Single-Pill Combination of Bisoprolol and Perindopril in Patients with Arterial Hypertension and Stable Coronary Artery Disease in Daily Clinical Practice: The STYLE Study. Adv Ther. 2021 Jun;38(6):3299-3313. doi: 10.1007/s12325-021-01754-2. Epub 2021 May 15. PMID 33991323

RESULTS

PARTICIPANT FLOW:
Groups:
- the Patients With HT and Concomitant Stable CAD: Observational study - 1 group - bisoprolol/perindopril FDC: single-pill combination of beta-blocker and ACE inhibitor
Period: Inclusion
Arm/Group | the Patients With HT and Concomitant Stable CAD
Started | 1909 (Planned to include 1920 pts, included 1909)
FVFP | 1909
Completed | 1909
Not Completed | 0
Period: 1 Month After Inclusion
Arm/Group | the Patients With HT and Concomitant Stable CAD
Started | 1909
1 Month After Inclusion | 1909
Completed | 1909
Not Completed | 0
Period: 3 Month After Inclusion
Arm/Group | the Patients With HT and Concomitant Stable CAD
Started | 1909
3 Month After Inclusion | 1909
Completed | 1892
Not Completed | 17

BASELINE CHARACTERISTICS:
Population: 1909 patients were included however 17 were excluded from the population analysed due to violation of inclusion creteria. Therefore full analysis set is 1892.
Arm/Group | the Patients With HT and Concomitant Stable CAD
Number analyzed (Participants) | 1892
Age, Categorical [Count of Participants; unit: Participants] — patients with arterial hypertension and stable coronary heart disease
  Participants
    <=18 years | 0
    Between 18 and 65 years | 1192
    >=65 years | 700
Sex: Female, Male [Count of Participants; unit: Participants] — Population: - in 11 participants no gender indicated
  Participants
    number analyzed (Participants) | 1881
    Female | 1007
    Male | 874
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 1909

OUTCOME MEASURES:

1. Primary Outcome: The Mean SBP Changes (mm Hg) at the Visit 3 vs. Baseline
Description: Changes in the mean office systolic BP levels (in mm Hg) in the sitting position
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Mean of SBP Changes: Changes in the mean office systolic BP levels (in mm Hg) in the sitting position among the patients with HT and CAD recieved the biso/perindopril FDC
Arm/Group | Mean of SBP Changes
Number analyzed (Participants) | 1892
mm Hg | 31.5 (14.2)

2. Primary Outcome: Efficacy of Bisoprolol/Perindopril FDC in Patients With HT and Stable CAD in Everyday Practice Regarding the BP: % of Patients Achieving Target Levels
Description: The percentage of the patients achieved the target levels of clinical BP among included patients ( SBP < 140 mm Hg and DBP < 90 mm Hg) with HT and stable CAD recieving Bisoprolol/Perindopril FDC
Time Frame: 3 month
Measure: Count of Participants; unit: Participants
Groups:
- the Patients With HT and Concomitant Stable CAD: Observational study - 1 group - bisoprolol/perindopril FDC: single-pill combination of beta-blocker and ACE inhibitor
  All patients included in the study received a FDC of beta-blocker bisoprolol and ACE inhibitor perindopril. In accordance with the investigation schedule, during the study the investigators collected subjective data from patients on the treatment compliance and tolerability (complaints), performed physical and instrumental examinations, as well as collected data from patients regarding the number of angina attacks and consumption of short-acting nitrates, adverse events/reactions, and assessed their quality of life using the visual analogue scale (VAS).
Arm/Group | the Patients With HT and Concomitant Stable CAD
Number analyzed (Participants) | 1892
Participants | 1640

3. Primary Outcome: Efficacy of Bisoprolol/Perindopril FDC in Patients With HT and Stable CAD in Everyday Practice: # of Angina Attacks
Description: Average decrease of the number of angina attacks in patients with HT and stable CAD who recieved the bisoprolol/perindopril FDC
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: number of angina attacks per week
Groups:
- the Patients With HT and Concomitant Stable CAD: the patients with HT and concomitant stable CAD recieved bisoprolol/perindopril FDC
Arm/Group | the Patients With HT and Concomitant Stable CAD
Number analyzed (Participants) | 1892
number of angina attacks per week | -3.2 (8.2)

4. Primary Outcome: Changes in the Mean Office Diastolic BP Levels (in mm Hg) in the Sitting Position
Description: Changes in the mean office diastolic BP levels (in mm Hg) in the sitting position among the patints with HT and CAD recieving bis/perindopril FDC
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Mean Office DBP Changes Between v3 vs Baseline: mean office DBP changes between v3 vs baseline among patients with HT and CAD recieving biso/perindopril FDC
Arm/Group | Mean Office DBP Changes Between v3 vs Baseline
Number analyzed (Participants) | 1892
mm Hg | 15.9 (9.5)

5. Secondary Outcome: Impact on the Quality of Life of Bisoprolol/Perindopril FDC in Patients With HT and Stable CAD in Everyday Practice: VAS
Description: Changes of the score in the visual analog scale (VAS) to assess the wellbeing; (minimum score 0 mm and maximum score 100 mm) among patients with HT and CAD recieving biso/perindopril FDC
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: units on a scale - mm
Arm/Group | the Patients With HT and Concomitant Stable CAD
Number analyzed (Participants) | 1892
units on a scale - mm | 35.1 (18.5)

6. Secondary Outcome: Good and Moderate Adherence to Bisoprolol/Perindopril FDC Therapy in Patients With HT and Stable CAD in Everyday Practice
Description: Percentage of the patients with definite answer on question from questionnaire regarding adherence; (Compliance evaluation test - 6 questions tes; Answer "No" to all questions: good compliance; Answer "Yes" to 1-2 questions: minor compliance; Answer "Yes" to 3 or more questions: noncompliance)
Time Frame: 3 month
Measure: Count of Participants; unit: Participants
Arm/Group | the Patients With HT and Concomitant Stable CAD
Number analyzed (Participants) | 1892
Participants | 1827

ADVERSE EVENTS:
Time Frame: 3 month
Description: Were registered 9 AEs in 4 patients, of which 3 patients had adverse drug reactions resulting in the withdrawal from treatment. 1 patient started to take the study drug periodically and not daily, which did not comply with the instructions for the medical use of the drug.
Arm/Group | the Patients With HT and Concomitant Stable CAD
All-Cause Mortality (participants affected / at risk) | 1/1909
Serious Adverse Events (participants affected / at risk) | 7/1909
Other Adverse Events (participants affected / at risk) | 2/1909
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | the Patients With HT and Concomitant Stable CAD (N=1909)
Non-traumatic vertebral compression fracture that required hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1)
death of unknown caus (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypotension with dizziness (Cardiac disorders) | 2 (2)
bradycardia (Product Issues) | 1 (1)
bradycardia (Cardiac disorders) | 1 (1)
syncope (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | the Patients With HT and Concomitant Stable CAD (N=1909)
Dry cough and tingling throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
A special situation: use of the drug not daily, but as needed (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03730116/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03730116/ICF_001.pdf